CLINICAL TRIAL: NCT01870388
Title: A Pharmacokinetic Study of Baricitinib in Subjects With Hepatic Dysfunction
Brief Title: A Pharmacokinetic Study of Baricitinib in Participants With Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14600; I4V-MC-JAGC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Liver Diseases; Hepatic Insufficiency
MeSH Terms: conditions — Liver Diseases; Hepatic Insufficiency | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baricitinib (Healthy) (Experimental): Group 1: 4 milligrams (mg) baricitinib administered once, orally, to participants with normal hepatic function.
  Interventions: Drug: Baricitinib
- Baricitinib (Moderate) (Experimental): Group 2: 4 mg baricitinib administered once, orally, to participants with moderate hepatic impairment.
  Interventions: Drug: Baricitinib
- Baricitinib (Mild) (Experimental): Group 3: 4 mg baricitinib administered once, orally, to participants with mild hepatic impairment. Enrollment is contingent on data from Groups 1 and 2.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104

SUMMARY:
The main purpose of this study is to measure how much of the study drug called baricitinib gets into the blood stream and how long it takes the body to get rid of it. Healthy participants and those with liver disease may enroll. The study will last about 7 days for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria for ALL Participants:

* Male participants agree to use 2 reliable methods of birth control with female partners of child-bearing potential during the study and for at least 3 months following the last dose of study drug
* Women not of child-bearing potential due to surgical sterilization (at least 6 weeks after surgical bilateral oophorectomy with or without hysterectomy or at least 6 weeks after confirmed tubal occlusion/tubal ligation) confirmed by medical history or menopause
* Menopausal women with spontaneous amenorrhea for at least 12 months, not induced by a medical condition and by medications and have a follicle-stimulating hormone (FSH) level greater than 40 milli-international units per milliliter (mIU/mL) (unless the participant is taking hormone replacement therapy [HRT])
* Have a body mass index of 18.5 to 40.0 kilograms per square meter (kg/m^2) inclusive at the time of screening

Additional Inclusion Criteria for Healthy Participants:

* Are overtly healthy participants, have normal hepatic function and have stable chronic medical conditions
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator

Additional Inclusion Criteria for Hepatically Impaired Participants:

* Participants with hepatic impairment classified as Child-Pugh score A or B (mild [Group 3, if enrolled] or moderate [Group 2] impairment, respectively). Must have a diagnosis of chronic hepatic impairment (greater than 6 months), with no clinically significant changes within 90 days prior to study drug administration (Day 1). Participants may have mild stable baseline medical conditions for which neither the condition nor treatments received would negatively impact the health of the participant or study conduct
* Clinical laboratory test results with deviations that are judged by the investigator to be compatible with the hepatic impairment of the participant, or of no additional clinical significance for this study

Exclusion Criteria for ALL Participants:

* Have received, within the last 30 days, an investigational product as part of a clinical trial, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Persons who have previously completed or withdrawn from study investigating baricitinib, and have previously received the investigational product
* Women with a positive pregnancy test or who are lactating
* Have a current or recent history (less than 30 days prior to screening and/or less than 45 days prior to admission to the clinical research unit) of a clinically significant bacterial, fungal, parasitic, viral (excluding rhinopharyngitis), or mycobacterial infection
* Have had symptomatic herpes zoster or herpes simplex infection within 90 days prior to the first dose
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Have been exposed to a live vaccine within 12 weeks prior to the first dose or expected to need/receive a live vaccine (including herpes zoster vaccination) during the course of the study

Additional Exclusion Criteria for Healthy Participants:

* Show evidence of acute or chronic liver disease
* Show evidence of hepatitis B and/or positive hepatitis B and/or positive hepatitis B surface antigen
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Intend to use over-the-counter or prescription medication and/or herbal supplements within 14 days prior to dosing and during the study

Additional Exclusion Criteria for Liver Impaired Participants:

* Have creatinine clearance less than or equal to 50 milliliter per minute (mL/min) using the Cockcroft and Gault formula
* Show evidence of spontaneous bacterial peritonitis within 6 month of dosing
* Have had variceal bleeding within 3 months of check in
* Show evidence of severe hyponatremia (sodium less than 120 millimolar per liter (mmol/L)
* Have severe encephalopathy (Grade 3 to 4)
* Have moderate to severe ascites (moderately hepatically impaired participants only)
* Show presence of a portal shunt
* Have hemoglobin less than 9.0 grams per deciliter (g/dL)
* Have serum bilirubin greater than 15 milligrams per deciliter (mg/dL)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An interim analysis was to be performed after ≤6 participants (pts) each in Group (G) 1 and G2 completed the study. If a <1.3-fold difference in exposure was seen between pts with moderate hepatic impairment (G2) and pts with normal hepatic function (G1), then pts with mild hepatic impairment (G3) were not to be enrolled. No pt was enrolled in G3.
Groups:
- Baricitinib (Healthy Participants): Group 1: A single 4-milligram (mg) dose of baricitinib (one 4-mg tablet) administered once, orally, to participants with normal hepatic function.
- Baricitinib (Moderate Hepatic Impairment): Group 2: A single 4-mg dose of baricitinib (one 4-mg tablet) administered once, orally, to participants with moderate hepatic impairment as classified by Child-Pugh B.
Period: Overall Study
Arm/Group | Baricitinib (Healthy Participants) | Baricitinib (Moderate Hepatic Impairment)
Started | 8 | 8
Received 1 Dose of Study Drug | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Baricitinib (Healthy Participants): Group 1: A single 4-mg dose of baricitinib (one 4-mg tablet) administered once, orally, to participants with normal hepatic function.
- Total: Total of all reporting groups
Arm/Group | Baricitinib (Healthy Participants) | Baricitinib (Moderate Hepatic Impairment) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Baricitinib (LY3009104)
Time Frame: Predose up to 48 hours (h) postdose
Population: Participants who received 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Baricitinib (Healthy Participants): Group 1: A single 4-mg dose of baricitinib (one 4-mg tablet) administered once, orally to participants with normal hepatic function.
- Baricitinib (Moderate Hepatic Impairment): Group 2: A single 4-mg dose of baricitinib (one 4-mg tablet) administered once, orally to participants with moderate hepatic impairment as classified by Child-Pugh B.
Arm/Group | Baricitinib (Healthy Participants) | Baricitinib (Moderate Hepatic Impairment)
Number analyzed (Participants) | 8 | 8
nanograms per milliliter (ng/mL) | 35.3 (25) | 38.2 (23)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity [AUC(0-∞)] of Baricitinib
Time Frame: Predose up to 48 h postdose
Population: Participants who received 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Baricitinib (Healthy Participants) | Baricitinib (Moderate Hepatic Impairment)
Number analyzed (Participants) | 8 | 8
nanograms*hour/milliliter (ng*h/mL) | 295 (25) | 350 (28)

ADVERSE EVENTS:
Arm/Group | Baricitinib (Healthy Participants) | Baricitinib (Moderate Hepatic Impairment)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib (Healthy Participants) (N=8) | Baricitinib (Moderate Hepatic Impairment) (N=8)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days